CLINICAL TRIAL: NCT02040792
Title: A Phase 2B, 28-Day, Randomized, Double-Blind Placebo-Controlled Parallel Group Study of Nebulized TD-4208 in Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: A 28-Day Parallel Group Study of TD-4208 in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0117
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: COPD
Keywords: COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — revefenacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 44 mcg (Experimental): TD-4208
  Interventions: Drug: TD-4208
- 88 mcg (Experimental): TD-4208
  Interventions: Drug: TD-4208
- 175 mcg (Experimental): TD-4208
  Interventions: Drug: TD-4208
- 350 mcg (Experimental): TD-4208
  Interventions: Drug: TD-4208

INTERVENTIONS:
Drug: TD-4208
  Other Names: revefenacin
  Arms: 175 mcg; 350 mcg; 44 mcg; 88 mcg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study evaluated the safety and efficacy of four doses of TD-4208 and a placebo product when administered once daily for 28 days using a jet nebulizer to patients with moderate to severe chronic obstructive pulmonary disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female subject 40 years of age or older
* Subject must have a negative pregnancy test, and must be prepared to use effective contraception if of child-bearing potential
* Subject is capable of performing reproducible spirometry maneuvers
* Subject has post-bronchodilator FEV1/FVC ratio <0.7
* Subject has moderate-to-severe stable COPD (Stage 2 or 3 according to the GOLD Guidelines)
* Subject has a post-bronchodilator FEV1 greater than or equal to 30% and less than 80% of predicted normal
* Subject has a current or past smoking history of at least 10 pack-years.

Exclusion Criteria:

* Subject has a significant respiratory disease or disorder other than COPD that would affect the interpretation of data from this study
* Subject has a history of reactions or hypersensitivity to inhaled or nebulized anticholinergic or beta-agonist agents
* Subject suffers from any medical condition that would preclude the use of inhaled anticholinergic agents
* Subject has been hospitalized for COPD or pneumonia within 12 weeks
* Subject requires long-term oxygen therapy (>15 hours a day)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medial Monitor, Study Director — Theravance Biopharma
Locations (1):
- Upstate Pharmaceutical Research, Greenville, South Carolina, United States

REFERENCES:
- [Derived] Lo A, Borin MT, Bourdet DL. Population Pharmacokinetics of Revefenacin in Patients with Chronic Obstructive Pulmonary Disease. Clin Pharmacokinet. 2021 Mar;60(3):391-401. doi: 10.1007/s40262-020-00938-3. PMID 33124005
- [Derived] Pudi KK, Barnes CN, Moran EJ, Haumann B, Kerwin E. A 28-day, randomized, double-blind, placebo-controlled, parallel group study of nebulized revefenacin in patients with chronic obstructive pulmonary disease. Respir Res. 2017 Nov 2;18(1):182. doi: 10.1186/s12931-017-0647-1. PMID 29096627

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject who received placebo was excluded from the efficacy analysis. The reason for this is that the subject was found to be participating in a GSK (GlaxoSmithKline) study with another investigational agent at the same time as their participation in this study.
Period: Overall Study
Arm/Group | Placebo | 44 mcg | 88 mcg | 175 mcg | 350 mcg
Started | 70 | 68 | 71 | 71 | 74
Completed | 64 | 65 | 68 | 64 | 67
Not Completed | 6 | 3 | 3 | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 44 mcg | 88 mcg | 175 mcg | 350 mcg | Total
Number analyzed (Participants) | 70 | 68 | 71 | 71 | 74 | 354
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (9.17) | 60.9 (8.87) | 60.4 (7.98) | 64.5 (7.69) | 61.4 (8.98) | 61.9 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 39 | 34 | 34 | 176
  Male | 37 | 32 | 32 | 37 | 40 | 178

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 (Forced Expiratory Volume in One Second)
Time Frame: Baseline to 28 days
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Placebo | 44 mcg | 88 mcg | 175 mcg | 350 mcg
Number analyzed (Participants) | 70 | 68 | 71 | 71 | 74
mL | -32.4 (25.36) | 19.4 (24.98) | 155.0 (24.61) | 134.2 (25.07) | 138.2 (24.38)

ADVERSE EVENTS:
Description: One subject who received placebo was excluded from the efficacy analysis. The reason for this is that the subject was found to be participating in a GSK study with another investigational agent at the same time as their participation in this study.
Arm/Group | Placebo | 44 mcg | 88 mcg | 175 mcg | 350 mcg
Serious Adverse Events (participants affected / at risk) | 0/71 | 1/68 | 0/71 | 2/71 | 1/74
Other Adverse Events (participants affected / at risk) | 8/71 | 1/68 | 6/71 | 10/71 | 15/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=71) | 44 mcg (N=68) | 88 mcg (N=71) | 175 mcg (N=71) | 350 mcg (N=74)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=71) | 44 mcg (N=68) | 88 mcg (N=71) | 175 mcg (N=71) | 350 mcg (N=74)
Headache (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
COPD (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Oropharyngeal pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may communicate the trial results generated by the PI, but only after the first publication or presentation of the combined study results generated by all participating sites. The Sponsor can then review trial results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days. The Sponsor cannot require changes to the communication and cannot extend the embargo.